CLINICAL TRIAL: NCT01191112
Title: Evaluation of the Safe Use and Tolerance of a Peptide-based Formula in a Pediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BK87
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Diseases; Feeding Intolerance
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peptide Based enteral formula (Experimental)
  Interventions: Other: Peptide based enteral formula

INTERVENTIONS:
Other: Peptide based enteral formula — Sole source nutrition as per HCP

SUMMARY:
The objective of this study is to determine the safe use and tolerance of a peptide-based formula in children with gastrointestinal dysfunction and/or feeding intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female between 1 and 13 years of age.
* Subject is diagnosed with gastrointestinal dysfunction and/or feeding intolerance.
* Subject requires enteral tube feeding as sole source of nutrition.

Exclusion Criteria:

* History of diabetes.
* Requires artificial ventilation.
* Requires parenteral nutrition.
* Subject has intestinal obstruction.
* Subject is receiving dialysis treatment.
* Subject has an allergy or intolerance to any ingredient in the study product.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 14 Days
Frequency and intensity of irritability, vomiting, distension | 14 Days

SECONDARY OUTCOMES:
Average Energy Intake | 14 Days
Anthropometrics | 14 Days
Medication Use | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MPH, Study Chair — Abbott Nutrition
Locations (1):
- University of Alberta, Stollery Children's Hospital, Edmonton, Alberta, Canada